CLINICAL TRIAL: NCT00866294
Title: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Clinical Effects of Controlled Release Paroxetine in the Treatment of Major Depressive Disorder
Brief Title: Controlled-release Paroxetine in Major Depressive Disorder (Double-blind, Placebo-controlled Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112810
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2010-11-15 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Depressive Disorder
Keywords: Immediate-release formulation of paroxetine (paroxetine IR); HAM-D (17 items); Controlled-release formulation of paroxetine (paroxetine CR)
MeSH Terms: conditions — Depressive Disorder | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- paroxetine CR group (Experimental): controlled-release (CR) of paroxetine 12.5 to 50mg/day
  Interventions: Drug: matched placebo to paroxetine IR 10mg or 20mg; Drug: Paroxetine CR 12.5mg tablet; Drug: Paroxetine CR 25mg tablet; Drug: matched placebo to paroxetine CR 12.5mg or 25mg
- paroxetine IR group (Other): Immediate-release (IR) of paroxetine 10 to 40mg/day as a reference arm
  Interventions: Drug: paroxetine IR 10mg tablet; Drug: paroxetine IR 20mg tablet; Drug: matched placebo to paroxetine IR 10mg or 20mg; Drug: matched placebo to paroxetine CR 12.5mg or 25mg
- placebo group (Placebo Comparator): matched placebo to both paroxetine CR and paroxetine IR
  Interventions: Drug: matched placebo to paroxetine IR 10mg or 20mg; Drug: matched placebo to paroxetine CR 12.5mg or 25mg

INTERVENTIONS:
Drug: paroxetine IR 10mg tablet — 1 or 2 tablets once a day
  Arms: paroxetine IR group
Drug: paroxetine IR 20mg tablet — 1 tablet once a day
  Arms: paroxetine IR group
Drug: matched placebo to paroxetine IR 10mg or 20mg — 1 or 2 tablets once a day
Drug: Paroxetine CR 12.5mg tablet — 1 or 2 tablets once a day
  Arms: paroxetine CR group
Drug: Paroxetine CR 25mg tablet — 1 or 2 tablets once a day
  Arms: paroxetine CR group
Drug: matched placebo to paroxetine CR 12.5mg or 25mg — 1 or 2 tablets once a day

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy of controlled-release (CR) formulation of paroxetine orally administered to patients with major depressive disorder (MDD) at a dose level in the range of 25 - 50 mg/day (initial dose level, 12.5 or 25 mg/day) once daily after evening meal for 8 weeks based on the decrease in HAM-D (Hamilton Depression Rating Scale) total score, to evaluate the safety based on adverse events, laboratory data and vital signs, and to describe the efficacy and safety of immediate release (IR) formulation of paroxetine.

ELIGIBILITY:
Inclusion Criteria:

<at the start of placebo run-in phase> Only the patients who meet all of the following conditions at Week -1 (at the start of placebo run-in phase) will be enrolled in this study. The hospitalization status will be no object. and Gender: No object.

* Target disease: Patients diagnosed as having one of the following depressive disorders based on DSM-IV-TR classification in conjunction with M.I.N.I. (The Mini International Neuropsychiatric Interview, Japanese version 5.0.0. [2003]) and showing currently a symptom of depression or depressed sate
* Major depressive disorder, single episode (296.2) (excluding those accompanied by comorbid psychiatric disorders)
* Major depressive disorder, recurrent (296.3) (excluding those accompanied by comorbid psychiatric disorders)
* Age: >= 20 years (at the time of obtaining consent)
* Consent: Patients from whom written consent to participate in this study can be obtained
* Gender:
* Female patients of childbearing potential can be enrolled. But, such patients who can be enrolled are limited to only those who are negative in the pregnancy test performed at the start of the placebo run-in phase and who agree to receive a pregnancy test at the time point defined in the study period and surely perform any of the contraceptive methods.
* Male subjects must abstain from (or use a condom during) sexual intercourse with a pregnant or lactating female. Male subjects must abstain from or use a condom plus spermicidal agent (foam/gel/film/cream/suppository) during sexual intercourse with a female of child-bearing potential.
* Patients whose HAM-D (17 items) total score is >= 20 points
* Patients whose duration of current episode at least 12 weeks but no longer than 24 months
* Patients whose score of "depressed mood" (HAM-D Item 1) is >= 2 points
* QTc<450 millisecond (msec) or <480 msec for patients with Bundle Branch Block - values based on either single ECG values or triplicate ECG averaged QTc values obtained over a brief recording period.

For the purposes of these criteria, QTc B (Bazett's correction) is defined as (QT interval [msec]) /(square root of RR interval [seconds])

<at the start of treatment phase> Only the patients who meet all of the following conditions at Week -1 (at the start of the placebo run-in phase) and Week 0 (at the start of treatment phase) can be shifted to the treatment phase.

* Patients whose HAM-D (17 items) total score is >=20 points
* Patients whose score of "depressed mood" (HAM-D Item 1) is >=2 points

Exclusion Criteria:

<at the start of placebo run-in phase> The patients who are meeting any of the following conditions at Week -1 (at the start of placebo run-in phase) must not be enrolled in this study.

* Patients whose primary diagnosis is a disorder classified to Axis I other than major depressive disorder in DSM-IV-TR classification (dysthymic disorder, eating disorder, specific phobia (monophobia), posttraumatic stress disorder, obsessive-compulsive disorder, panic disorder, etc.)
* Patients with a current DSM-IV-TR Axis II diagnosis that suggested non-responsiveness to pharmacotherapy or non- compliance with the protocol (e.g., antisocial or borderline personality disorder)
* Patients with a history or complication of another (non-MDD) mental disorder (schizophrenia, etc.)
* Patients with a history or complication of manic episodes
* Patients diagnosed as having an attentional deficit disorder or hyperactivity disorder
* Patients diagnosed as having a pervasive development disorder or mental retardation
* Patients diagnosed as abusing or dependent on alcohol or drug within one year before the Week -1 visit
* Patients who have undergone electroconvulsive therapy within one year before the Week -1 visit for the treatment of the current episode
* Patients who have a history of treatment with depot neuroleptics
* Patients with a history of serotonin syndrome or neuroleptic malignant syndrome
* Patients with a >= 3-point score of "suicide" (HAM-D Item 3) or patients whose Columbia Suicide Severity Rating Scale (C-SSRS) assessment suggests that they are or have been at significant risk for harming themselves or have actually harmed themselves, or who, in the opinion of the investigator (subinvestigator), are at significant risk for harming self or others.
* Patients with a history of suicide attempt, self-injurious action (excluding action with no intention of suicide) or overdosage (excluding apparently accidental overdosage)
* Patients who have taken another investigational product or a drug used in a post-marketing clinical study within 12 weeks before the Week -1 visit
* Patients with glaucoma
* Patients with a convulsive disorder such as epilepsy or a history of it
* Patients using a drug increasing an onset risk of bleeding, patients with a bleeding tendency or bleeding diathesis
* Patients complicated with severe renal or hepatic dysfunction
* Patients complicated with serious organic brain disorder
* Patients with a history or complication of cancer or malignant tumor
* Patients complicated by chronic hepatitis B or C being positive in test of hepatitis B surface antigen (HbsAg) or hepatitis C antibody
* Pregnant, lactating or possibly pregnant female patients, and female patients wishing to be pregnant during the study period
* Patients who have previously been unresponsive to paroxetine therapy (e.g. >4wks unresponsive to paroxetine for depression).
* Patients with a history of having discontinued treatment due to an adverse event caused by paroxetine
* Patients with a history of hypersensitivity to paroxetine.
* Patients judged ineligible to participate in this study by the investigator or subinvestigator

Exclusion criteria < at the start of treatment phase> The patients who are meeting any of the following conditions at Week 0 (at the start of treatment phase) must not be allowed to the treatment phase.

* Patients with a 3 or more-point score of "suicide" (HAM-D Item 3) or with a strong suicidal tendency by C-SSRS and investigator clinical judgement.
* Patients whose HAM-D (17 items) total score at the Week 0 visit has changed ±25 %, or exceeding the range of ±25 % of the score at the Week -1 visit
* Patients whose Drug 1 (run-in placebo) compliance rate in the period from Week -1 to Week 0 has been < 80 %
* Patients judged ineligible as the study subjects by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- Japan (17):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
- South Korea (2):
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Higuchi T, Hong JP, Jung HY, Watanabe Y, Kunitomi T, Kamijima K. Paroxetine controlled-release formulation in the treatment of major depressive disorder: a randomized, double-blind, placebo-controlled study in Japan and Korea. Psychiatry Clin Neurosci. 2011 Dec;65(7):655-63. doi: 10.1111/j.1440-1819.2011.02243.x. Epub 2011 Sep 6. PMID 21895859
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had completed all the study procedures (up to the post-study examinations) were defined as per protocol completers.
Groups:
- Placebo: Placebo matched to the controlled release formulation (CR) of paroxetine and placebo matched to the immediate release formulation (IR) of paroxetine were administered orally once daily from the start of the treatment phase (8 weeks) through the end of the taper phase (0-3 weeks).
- Paroxetine CR: An initial dose of 12.5 or 25 milligrams (mg)/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Thereafter, 25-50 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 12.5 mg/day were forced to receive the uptitrated dose of 25 mg/day, and participants who started the treatment from 25 mg/day were maintained at the same dose level. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 12.5 mg/day at weekly intervals to the final dose level of 12.5 mg/day to complete the treatment.
- Paroxetine IR: An initial dose of 10 or 20 mg/day of paroxetine IR was administered orally once daily in the first week of the treatment phase. Thereafter, 20-40 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 10 mg/day were forced to receive the uptitrated dose of 20 mg/day, and participants who started the treatment from 20 mg/day were maintained at the same dose level. The dose level was increased by 10 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 10 mg/day at weekly intervals to the final dose level of 10 mg/day to complete the treatment.
Period: Overall Study
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Started | 172 | 161 | 83
Completed | 139 | 141 | 72
Not Completed | 33 | 20 | 11
Not completed — Adverse Event | 12 | 13 | 9
Not completed — Lack of Efficacy | 7 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Met Protocol-defined Stopping Criteria | 5 | 1 | 1
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Physician Decision | 6 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR | Total
Number analyzed (Participants) | 172 | 161 | 83 | 416
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (10.04) | 36.4 (11.36) | 35.5 (10.38) | 36.4 (10.62)
Gender [Count of Participants; unit: Participants]
  Female | 94 | 86 | 48 | 228
  Male | 78 | 75 | 35 | 188
Race/Ethnicity, Customized [Number; unit: participants] — The number of participants is based on the Full Analysis Set (FAS), consisting of all participants who entered the treatment phase, excluding those who had taken no dose of the investigational product for the treatment phase and those who had no data on the Hamilton Depression Rating Scale (HAM-D) total score after the start of the treatment phase.
  participants
    Asian - East Asian Heritage | 17 | 20 | 10 | 47
    Asian - Japanese Heritage | 154 | 138 | 73 | 365

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in the Hamilton Depression Rating Scale (HAM-D; 17 Items) Total Score at Week 8
Description: The HAM-D measures the severity of depressive symptoms in participants with major depressive disorder (MDD). It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms. Mean change from baseline was calculated as the value at Week 8 minus the Baseline value.
Time Frame: Baseline (Week 0) and Week 8
Population: Full Analysis Set (FAS): all participants who entered the treatment phase (8 weeks), excluding those who had taken no dose of the investigational product for the treatment phase and who had no data on the HAM-D total score after the start of the treatment phase. The analysis was performed on the last observation carried forward (LOCF) dataset.
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo: Placebo matched to the controlled release formulation (CR) of paroxetine and placebo matched to the immediate release formulation (IR) of paroxetine were administered orally once daily.
- Paroxetine CR: An initial dose of 12.5 or 25 milligrams (mg)/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Thereafter, 25-50 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 12.5 mg/day were forced to receive the uptitrated dose of 25 mg/day, and participants who started the treatment from 25 mg/day were maintained at the same dose level. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed.
- Paroxetine IR: An initial dose of 10 or 20 mg/day of paroxetine IR was administered orally once daily in the first week of the treatment phase. Thereafter, 20-40 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 10 mg/day were forced to receive the uptitrated dose of 20 mg/day, and participants who started the treatment from 20 mg/day were maintained at the same dose level. The dose level was increased by 10 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed.
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
scores on a scale | -10.4 (0.62) | -12.8 (0.61) | -12.5 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Paroxetine CR; Test type: Superiority or Other; p < 0.001, ANCOVA — The hypothesis test was conducted with a two-sided significance level of 5% to show the superiority of paroxetine CR relative to placebo; The primary analysis was based on an ANCOVA with a model adjusting for baseline HAM-D total score and region (Japan and South Korea); Mean Difference (Net) = -2.4, 95% CI 2-sided [-3.8 to -1.1] — Mean difference = paroxetine CR minus placebo

2. Secondary Outcome: Mean Change From Baseline in the HAM-D Total Score at Weeks 1, 2, 3, 4, 6, and 8
Description: The HAM-D measures the severity of depressive symptoms in participants with MDD. It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms. Mean change from baseline was calculated as the value at each time point minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 1, 2, 3, 4, 6, and 8
Population: FAS. The analysis was performed on the following datasets: the observed case (OC) dataset for Week 1 and the LOCF dataset for Weeks 2, 3, 4, 6, and 8, where missing values were imputed by the last observed value in the longitudinal data. One participant in the Paroxetine CR group was not included in the OC analysis for having a missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo: Placebo matched to paroxetine CR and placebo matched to paroxetine IR were administered orally once daily.
- Paroxetine CR: An initial dose of 12.5 or 25 mg/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Thereafter 25-50 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 12.5 mg/day were forced to receive the uptitrated dose of 25 mg/day and participants who started the treatment from 25 mg/day were maintained at the same dose level. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed.
- Paroxetine IR: An initial dose of 10 or 20 mg/day of paroxetine IR was administered orally once daily in the first week of the treatment phase. Thereafter 20-40 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 10 mg/day were forced to receive the uptitrated dose of 20 mg/day and participants who started the treatment from 20 mg/day were maintained at the same dose level. The dose level was increased by 10 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed.
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
scores on a scale
  Week 1, n=171, 157, 83 | -3.1 (4.04) | -2.9 (4.05) | -3.5 (4.36)
  Week 2, n=171, 158, 83 | -5.2 (5.11) | -5.5 (4.85) | -6.2 (4.93)
  Week 3, n=171, 158, 83 | -6.7 (6.05) | -7.5 (5.64) | -7.3 (4.70)
  Week 4, n=171, 158, 83 | -8.0 (6.10) | -9.3 (5.66) | -9.1 (5.66)
  Week 6, n=171, 158, 83 | -8.8 (6.40) | -10.9 (6.21) | -10.4 (5.78)
  Week 8, n=171, 158, 83 | -9.8 (6.68) | -12.4 (6.41) | -12.0 (5.83)

3. Secondary Outcome: Percentage of HAM-D Responders at Weeks 4 and 8
Description: The HAM-D measures the severity of depressive symptoms in participants with MDD. It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is a sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms. Responders are defined as participants with a 50 percent or greater reduction from baseline in the HAM-D total score.
Time Frame: Weeks 4 and 8
Population: FAS. The analysis was performed on the OC dataset. The analysis of Week 8 data was also performed on the LOCF dataset, where missing values were imputed by the last observed value in the longitudinal data. Some participants in each group were not included in the OC analysis because they were withdrawn prematurely.
Measure: Number; unit: percentage of responders
Groups:
- Paroxetine CR: An initial dose of 12.5 or 25 mg/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Thereafter, 25-50 mg/day was administered once daily for 7 weeks. In the second week, participants who started the treatment from 12.5 mg/day were forced to receive the uptitrated dose of 25 mg/day, and participants who started the treatment from 25 mg/day were maintained at the same dose level. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed.
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
percentage of responders
  Week 4, n=158, 154, 78 | 30 | 40 | 40
  Week 8 (OC), n=144, 145, 74 | 52 | 66 | 59
  Week 8 LOCF, n=171, 158, 83 | 46 | 63 | 57

4. Secondary Outcome: Percentage of HAM-D Remitters at Weeks 4 and 8
Description: The HAM-D measures the severity of depressive symptoms in participants with MDD. It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms. Remitters are defined as participants with a HAM-D total score of 7 or less.
Time Frame: Weeks 4 and 8
Population: as for outcome 3
Measure: Number; unit: percentage of remitters
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
percentage of remitters
  Week 4, n=158, 154, 78 | 16 | 15 | 18
  Week 8 (OC), n=144, 145, 74 | 26 | 38 | 39
  Week 8 LOCF, n=171, 158, 83 | 23 | 35 | 36

5. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-SI) Scores at Weeks 1, 2, 3, 4, 6, and 8
Description: The 7-point CGI-SI scale assesses the clinician's impression of the participant's current illness state. Scores on the CGI-SI range from 1 = not ill at all to 7 = among the most extremely ill. Mean change from baseline was calculated as the value at each time point minus the baseline value.
Time Frame: Baseline (Week 0); Weeks 1, 2, 3, 4, 6, and 8
Population: FAS. The analysis was performed on the OC dataset. The analysis of Week 8 data was also performed on the LOCF dataset, where missing values were imputed by the last observed value in the longitudinal data. Some participants in each group were not included in the OC analysis because they had missing values or they were withdrawn prematurely.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
scores on a scale
  Week 1, n=171, 157, 83 | -0.1 (0.46) | -0.2 (0.43) | -0.2 (0.58)
  Week 2, n=164, 155, 80 | -0.4 (0.68) | -0.4 (0.59) | -0.5 (0.67)
  Week 3, n=161, 155, 78 | -0.6 (0.83) | -0.7 (0.74) | -0.6 (0.72)
  Week 4, n=158, 153, 79 | -0.7 (0.85) | -0.8 (0.85) | -0.8 (0.93)
  Week 6, n=151, 147, 76 | -0.9 (0.87) | -1.1 (0.98) | -0.9 (0.90)
  Week 8, n=144, 145, 74 | -1.0 (0.96) | -1.3 (1.02) | -1.3 (1.01)
  Week 8 LOCF, n=171, 158, 83 | -0.9 (1.02) | -1.2 (1.02) | -1.1 (1.05)

6. Secondary Outcome: Percentage of Responders Based on the Clinical Global Impression-Global Improvement (CGI-GI) Scores at Weeks 4 and 8
Description: The 7-point CGI-GI assesses the participant's improvement or worsening from baseline. Scores on the CGI-GI range from 1 = very much improved to 7 = very much worse. Responders are defined as participants with a score of 1 or 2 = much improved.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Paroxetine CR | Paroxetine IR
Number analyzed (Participants) | 171 | 158 | 83
percentage of responders
  Week 4, n=158, 153, 79 | 40 | 51 | 56
  Week 8 (OC), n=144, 145, 74 | 60 | 76 | 78
  Week 8 LOCF, n=171, 158, 83 | 53 | 71 | 75

ADVERSE EVENTS:
Time Frame: AEs were collected from run-in (Week -1) through the end of the follow-up phase (up to Week 13). SAEs were collected from the time a participant consented to participate in the study up to and including any follow-up contact.
Groups:
- Placebo: Placebo matched to paroxetine CR and placebo matched to paroxetine IR were administered orally once daily from the start of the treatment phase (8 weeks) through the end of the taper phase (0-3 weeks).
- Paroxetine CR 12.5-50 mg/Day: An initial dose of 12.5 mg/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Then the dose was uptitrated to 25 mg/day, and 25-50 mg/day was administered once daily for 7 weeks. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 12.5 mg/day at weekly intervals to the final dose level of 12.5 mg/day to complete the treatment.
- Paroxetine CR 25-50 mg/Day: An initial dose of 25 mg/day of paroxetine CR was administered orally once daily in the first week of the treatment phase. Thereafter, 25-50 mg/day was administered once daily for 7 weeks. The dose level was increased by 12.5 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 12.5 mg/day at weekly intervals to the final dose level of 12.5 mg/day to complete the treatment.
- Paroxetine CR, Total: All participants receiving either paroxetine CR 12.5-50 mg/day or 25-50 mg/day
- Paroxetine IR 10-40 mg/Day: An initial dose of 10 mg/day of paroxetine IR was administered orally once daily in the first week of the treatment phase. Then the dose was uptitrated to 20 mg/day, and 20-40 mg/day was administered once daily for 7 weeks. The dose level was increased by 10 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 10 mg/day at weekly intervals to the final dose level of 10 mg/day to complete the treatment.
- Paroxetine IR 20-40 mg/Day: An initial dose of 20 mg/day of paroxetine IR was administered orally once daily in the first week of the treatment phase. Thereafter, 20-40 mg/day was administered once daily for 7 weeks. The dose level was increased by 10 mg/day at intervals of at least 1 week until sufficient efficacy was confirmed. During the taper phase, the last dose level in the treatment phase was reduced by 10 mg/day at weekly intervals to the final dose level of 10 mg/day to complete the treatment.
- Paroxetine IR, Total: All participants receiving either paroxetine IR 10-40 mg/day or 20-40 mg/day
Arm/Group | Placebo | Paroxetine CR 12.5-50 mg/Day | Paroxetine CR 25-50 mg/Day | Paroxetine CR, Total | Paroxetine IR 10-40 mg/Day | Paroxetine IR 20-40 mg/Day | Paroxetine IR, Total
Serious Adverse Events (participants affected / at risk) | 1/172 | 2/79 | 4/82 | 6/161 | 2/43 | 0/40 | 2/83
Other Adverse Events (participants affected / at risk) | 76/172 | 43/79 | 50/82 | 93/161 | 23/43 | 21/40 | 44/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Paroxetine CR 12.5-50 mg/Day (N=79) | Paroxetine CR 25-50 mg/Day (N=82) | Paroxetine CR, Total (N=161) | Paroxetine IR 10-40 mg/Day (N=43) | Paroxetine IR 20-40 mg/Day (N=40) | Paroxetine IR, Total (N=83)
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Paroxetine CR 12.5-50 mg/Day (N=79) | Paroxetine CR 25-50 mg/Day (N=82) | Paroxetine CR, Total (N=161) | Paroxetine IR 10-40 mg/Day (N=43) | Paroxetine IR 20-40 mg/Day (N=40) | Paroxetine IR, Total (N=83)
Nausea (Gastrointestinal disorders) | 14 | 8 | 21 | 29 | 8 | 8 | 16
Constipation (Gastrointestinal disorders) | 5 | 9 | 8 | 17 | 4 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 1 | 6 | 7 | 4 | 4 | 8
Dry mouth (Gastrointestinal disorders) | 7 | 3 | 4 | 7 | 2 | 3 | 5
Headache (Nervous system disorders) | 18 | 5 | 7 | 12 | 2 | 2 | 4
Somnolence (Nervous system disorders) | 4 | 11 | 5 | 16 | 4 | 3 | 7
Dizziness (Nervous system disorders) | 4 | 5 | 6 | 11 | 3 | 1 | 4
Tremor (Nervous system disorders) | 0 | 3 | 1 | 4 | 2 | 3 | 5
Nasopharyngitis (Infections and infestations) | 33 | 8 | 13 | 21 | 4 | 4 | 8
Withdrawal syndrome (Psychiatric disorders) | 10 | 12 | 17 | 29 | 3 | 2 | 5
Pollakiuria (Renal and urinary disorders) | 3 | 1 | 1 | 2 | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.